CLINICAL TRIAL: NCT01643148
Title: Phase 1. Collect Samples of Breast Biopsy Patients Treated at the Hospital Radiology Service Maternal Perinatal Monica Pretelini
Brief Title: The Tetrad BMI, Leptin, Leptin/Adiponectin (L/A) Ratio and CA-15-3 is a Reliable Biomarker of Breast Cancer
Acronym: leptin
Status: Completed | Type: Observational
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Collaborators: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, PhD, Materno-Perinatal Hospital of the State of Mexico
Other Study IDs: DCQ
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Female Breast Carcinoma
Keywords: biomarker; BMI; breast cancer; CA-15-3; leptin
MeSH Terms: conditions — Breast Neoplasms; Medullary cystic kidney disease 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- breast cancer patients (cases): 36 subjects
- controls: 36 subjects

SUMMARY:
Objective:

Evaluate body mass index (BMI), leptin, Leptin/adiponectin (L/A) ratio and cancer antigen (CA) 15-3 together as reliable biomarkers for breast cancer.

Patients:

Consecutive patients aged between 40 - 60 years, with breast disease and informed consent.

Interventions:

Patients' Anthropometric and laboratorial characteristics classified by BMI in the group of cancer and patients with benign breast disease as well as biochemical tests of leptin, adiponectin,CA 15-3, hemoglobin, glucose low-density lipoprotein cholesterol (LDLC), high-density lipoprotein cholesterol (HDLC) levels were obtained as well as a blood sample to analyze CA 15-3 levels with a electrochemiluminescence immunoassay.

Hypothesis:

Using together leptin, L/A ratio, CA 15-3 and BMI could offer a reliable approach to detect high risk women to develop breast cancer.

DETAILED DESCRIPTION:
Serum levels of leptin, adiponectin and CA 15-3, as well as anthropometric and biochemical parameters were analyzed in 88 female patients attending mammography study. Predictive values of BMI, leptin, L/A ratio and CA 15-3 were determined with 95% confidence interval (CI).

ELIGIBILITY:
Inclusion Criteria:

* Female patients attending mammography, average age of the fourth and fifth decades.

Exclusion Criteria:

* Patients with hormonal therapy.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cross-sectional prospective study conducted at the Maternal-Perinatal Hospital "Mónica Pretelini" (HMPMP), State of Mexico Health Institute (ISEM), Toluca, Mexico, from January to October 2011.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonnathan Guadalupe Santillán Benítez, MSc, Principal Investigator — Autonomus University Of the State Of México; Leobardo Manuel Gómez Oliván, PhD, Study Director — Universidad Autonoma del Estado de Mexico; Hugo Mendieta Zeron, PhD, Study Chair — Autonomous University of the State of Mexico

REFERENCES:
- [Derived] Santillan-Benitez JG, Mendieta-Zeron H, Gomez-Olivan LM, Torres-Juarez JJ, Gonzalez-Banales JM, Hernandez-Pena LV, Ordonez-Quiroz A. The tetrad BMI, leptin, leptin/adiponectin (L/A) ratio and CA 15-3 are reliable biomarkers of breast cancer. J Clin Lab Anal. 2013 Jan;27(1):12-20. doi: 10.1002/jcla.21555. Epub 2013 Jan 4. PMID 23292756